CLINICAL TRIAL: NCT04014452
Title: Microwave Ablation Versus Radiofrequency Ablation for the Treatment of Severe Complicated Monochorionic Pregnancies in the Peking University Third Hospital : A Pilot Randomised Controlled Trial
Brief Title: Microwave Ablation vs Radiofrequency Ablation in the Management of Complicated Monochorionic Pregnancies：A RCT Study
Acronym: MWAvsRFA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PekingUTHweiyuanRCT
Record Dates: First submitted 2019-06-22; First posted 2019-07-10 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Twin; Complicating Pregnancy; Microwave Ablation
Keywords: Complicated Monochorionic Pregnancies; Selective feticide
MeSH Terms: conditions — Pregnancy Complications | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician will seal the randomisation codes in sequentially numbered opaque envelopes and send them to the research centres. Allocation will be concealed until participants sign the informed consent, at which time the interventionalist will access the allocation code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microwave ablation group (Experimental): Microwave ablation is used for the treatment of Complicated Monochorionic Pregnancies
  Interventions: Procedure: Microwave ablation
- Radiofrequency ablation group (Active Comparator): Radiofrequency ablation is used for the treatment of Complicated Monochorionic Pregnancies
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Microwave ablation — Use of microwave energy to ablate tissue surrounding fetal umbilical cord. All the procedures are performed percutaneously under ultrasound guidance.
  Arms: Microwave ablation group
Procedure: Radiofrequency ablation — Use of radiofrequency energy to ablate tissue surrounding fetal umbilical cord. All the procedures are performed percutaneously under ultrasound guidance.
  Arms: Radiofrequency ablation group

SUMMARY:
Complicated pregnancies refer some special complications, including twin to twin transfusion syndrome(TTTS), twin reverse arterial perfusion(TRAP), selective intrauterine fetal growth restriction(sIUGR), twin anemia-polycythemia sequence(TAPS), one fetal death or structural abnormalities, etc. Complicated twins are often associated with high perinatal morbidity and mortality. Severe complicated twins can be treated with fetal-reduction surgery during pregnancy, which can improve the survival rate of retained fetuses and reduce the disability rate. The managements include mechanical umbilical cord ligation or thermal coagulation obliteration, such as bipolar coagulation (BCC), radiofrequency ablation (RFA), and laser coagulation.Nowadays radiofrequency ablation reduction is the most common, which processes a higher survival rate and fewer maternal and fetal complications compared with other ways.Latest experience suggests that microwave ablation(MWA) is also easy to be used and the therapeutic effect is similar with RFA, but there is no convincing evidence. Compared with radiofrequency ablation, MWA has the advantages of simple operation and time, and avoids the problems of tissue carbonization, drying and heat sink effect. For fetation reduction surgery, the main advantage is that the endothermic effect near the blood vessels is smaller, which enables microwave fetation reduction to have a larger ablation range and a higher thermal effect. This study is comparing Microwave Ablation(MWA) and radiofrequency ablation (RFA) methods for selective fetal reduction in the treatment of complicated monochorionic (MC) multifetal gestations.

This is a pilot randomised controlled trial(RCT) of 60 patients who undergo selective fetal reduction. The subjects of this study were all pregnant women and their offspring who underwent reduction surgery in the third hospital of Beijing University, and patients are randomly assigned 1:1 to different intervention groups by parallel design. The outcome evaluators were blind. Collecting their surgery, clinical information and maternal and fetal complications at a week and a month after surgery, 42 days and 6 months after delivery, to verify the safety and efficacy of MWA, and find a better treatment plan for complicated monochorionic pregnancies .The primary outcome was neonatal survival rate.

DETAILED DESCRIPTION:
Medical charts were reviewed for the details of surgery and the pregnancy outcomes if the patient delivered at the authors'institution. In the event of delivery at distant locations, patients were contacted by telephone to obtain delivery and neonatal information. Patients are randomly assigned 1:1 to different intervention groups by parallel design. Chorionicity was assessed by the referring physicians during the ﬁrst trimester. All patients underwent comprehensive ultrasound examination to confirm the fetal diagnosis, chorionicity, amnionicity and cervical length upon arrival at Peking University Third Hospital. Monochorionicity was confirmed through the ultrasound findings of a single placenta, a thin intervening membrane, lack of a lambda sign and concordance for fetal gender. Patients were counseled about the risks and benefits of expectant management vs. selective reduction. Written informed consent was obtained. Statistical analysis was performed using the statistical software Statistical Product and Service Solutions(SPSS), for comparison of entry and outcome variables using the chi-square test, Fisher's exact test and the Student's t-test, where appropriate. P < 0.05 was considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Complicated monochorionic pregnancies women;
2. Having the indication of selective reduction;(TTTS III or IV, TRAP, severe sIUGR, Twin malformation inconsistency or stillbirth，three or more fetuses with monochorionic pregnancies requiring reducing the number of fetuses）
3. The reduction surgery should be done after 15 weeks of gestation;
4. Willingness to participate in the trial and having provided written consent.

Exclusion Criteria:

1. Preoperative examination shows that patient is not appropriate to undergoing reduction surgery, such as acute infection of the organ system, especially the urinary system.
2. Patients need to perform acute reduction surgery due to the progress of the disease and the surgery cannot be scheduled.
3. Other diseases that may affect the experimental results: neuropsychiatric diseases and congenital diseases.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Neonatal survival rate | a month after delivery
  The proportion of live births at 28 days postpartum

SECONDARY OUTCOMES:
Surgical injury to fetal | at 28 weeks gestation
  Using MRI to assess postoperative thermal injury and nerve injury of fetus
Postoperative complications | at delivery
  Frequency of PPROM, premature delivery, frequency of infection, procedure-to-delivery interval, <28 weeks of intrauterine fetal death/abortion, >28 weeks of intrauterine fetal deat and <32 weeks premature delivery
Perinatal outcomes | a week after delivery
  Using Apgar Score to assess neonatal asphyxia（Heart rate, respiration, muscle tone, laryngeal reflex and skin color within one minute after birth are taken as the basis, each item is 0~2 points, the full mark is 10 points. 8~10 belong to normal newborns. 4~7 can be classified as mild asphyxiation, 0~3 as severe asphyxiation）
Growth of the children | 6 months postpartum
  The height of the surviving fetus at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Zeng Lin, Ph.D, Study Chair — PRS administrator
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Requested data for public purpose or research transparency will be provided via the corresponding author. Participant data after deidentification (text, table, figures, and appendices) and protocol will be shared beginning 9 months and ending 36 months following article publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Participant data after deidentification (text, table, figures, and appendices) and protocol will be shared beginning 9 months and ending 36 months following article publication
Access Criteria: Requested data for public purpose or research transparency will be provided via the corresponding author.The e-mail address is weiyuanbysy@163.com.

REFERENCES:
- [Derived] Xie J, Cheng Z, Wu T, Wei Y, Wang X. Microwave ablation versus radiofrequency ablation for the treatment of severe complicated monochorionic pregnancies in China：protocol for a pilot randomised controlled trial. BMJ Open. 2020 Aug 13;10(8):e034995. doi: 10.1136/bmjopen-2019-034995. PMID 32792427